CLINICAL TRIAL: NCT03374150
Title: The Effect of Diet Counseling for Low Calorie-High Protein on the Body Composition (Weight, Body Mass Index, Fat Mass (kg), Fat Mass Percentage, Muscle Mass (kg), Muscle Mass Percentage, Inflammation Marker (High-sensitivity C-reactive Protein), and Oxidative Stress Marker (Malondialdehyde and Glutathione) in Obese People With Weight Cycling in Jakarta
Brief Title: The Effect of Diet Counseling for Low Calorie-High Protein on the Body Composition, Inflammation Marker, and Oxidative Stress Marker in Obese People With Weight Cycling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Fiastuti Witjaksono, Principal Invdstigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PITTAgizi
Record Dates: First submitted 2017-12-03; First posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Low-Calorie Diet; Diet, High-Protein; Obesity; Pituitary; Weight Cycling
Keywords: Low-Calorie Diet; Diet, High-Protein; Obesity; weight cycling; body composition; high-sensitivity C-Reactive protein; malondialdehyde; glutathione
MeSH Terms: conditions — Obesity; Pituitary Diseases; Weight Cycling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high protein (Experimental): High protein (HP) group were given counseling about weight loss program by applying low calorie-high protein diet with diet menu composition of 22-30% protein, along with instructions for allowed cooking method.
  Interventions: Behavioral: diet counseling
- standard protein (Active Comparator): Active comparator receiving standard protein (SP) proportion were counseled about weight loss program by means of low calorie-balanced composition diet with menu comprised of 12-20% protein.
  Interventions: Behavioral: diet counseling

INTERVENTIONS:
Behavioral: diet counseling — Subjects were given nutrition consultation, diet recipes, and logbook. Counseling was performed once weekly. During 8 weeks of diet program, subjects were instructed to reduce their daily caloric intake by 500 - 1000 kcal from their previous usual daily intake with limitation in low calorie diet range (800-1500 kcal.day) of calorie intake.Follow-up for each subject was performed once daily by person-to-person encounter. Besides, subjects were contacted by everyday cellphone texting and telephone twice a week to control subject's compliance. After 8 weeks of intervention, subjects were invited to revisit the clinic for anthropometry and body composition measurement after completing the program.

SUMMARY:
The world prevalence of obesity in adult population in 2014 was nearly 13% while in Indonesia, it has reached 32.9% in the same year. Obesity is an established risk factors for cardiovascular diseases. A large proportion of people who had succeeded to reduce body weight failed to maintain it (weight cycling). Studies were inconclusive about the best composition in the diet for such people to have a better life quality and reduce risk factors from non-communicable disease. The purpose of this research was to evaluate the body composition changes, Inflammation marker and oxidative stress marker changes resulted from low calorie high protein and standard protein diet programme in obese people with history of weight cycling.

This is an open-randomized clinical trial of weight loss program as a part of a larger study researching the effect of low calorie high protein diet to body composition, oxidative stress, inflammation marker and metabolic syndrome in obese with weight cycling. Subjects were assigned to low calorie diet and were randomly distributed into two intervention groups, namely high protein group (22-30 % of total calories intake) and standard protein group (12-20%). Anthropometry, body composition data, and blood sample (for inflammation marker (HsCRP) and oxidative stress (malondialdehyde and glutathione)) were taken at baseline and at the end of the study. Subjects were followed up to 8 weeks with daily reminder and weekly counselling

ELIGIBILITY:
Inclusion Criteria:

* body mass index ranging from 25 - 35 kg/m2
* history of weight loss ≥2 kg and regaining weight into or exceeding its initial body weight at least twice in last five years

Exclusion Criteria:

* diabetes mellitus
* history of gastrointestinal tract resection
* hormonal disorders
* using hormonal contraception
* menopause,
* kidney function disruption

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2017-05-26 (Actual); Primary Completion 2017-12-14 (Estimated); Study Completion 2017-12-14 (Estimated)

PRIMARY OUTCOMES:
body weight | eight weeks
  body weight analyzed by body composition monitors with advanced bioelectrical impedance analysis (BIA) principle expressed in kilogram (kg) unit
body mass index | eight weeks
  a weight-to-height ratio, calculated by dividing one's weight in kilograms by the square of one's height in meters analyzed by body composition monitors with advanced bioelectrical impedance analysis (BIA) principle expressed in kilogram per meter squared (kg/m^2) unit
fat mass | eight weeks
  actual weight of fat in one's body analyzed by body composition monitors with advanced bioelectrical impedance analysis (BIA) principle expressed in kilogram (kg) unit
fat mass percentage | eight weeks
  the proportion of fat to the total body weight analyzed by body composition monitors with advanced bioelectrical impedance analysis (BIA) principle expressed as percentage (%)
muscle mass | eight weeks
  The predicted weight of muscle in one's body analyzed by body composition monitors with advanced bioelectrical impedance analysis (BIA) principle expressed in kilogram (kg) unit
muscle mass percentage | eight weeks
  The predicted proportion of muscle weight to the total body weight analyzed by body composition monitors with advanced bioelectrical impedance analysis (BIA) principle expressed in kilogram (kg) unit
Inflammation marker (high-sensitivity C-reactive protein) | eight weeks
  indicator of inflammation state measured by Immunochemiluminescent (Immulite 1000) device
plasma malondialdehyde level | eight weeks
  the concentration of malondialdehyde (1,3-Propanedial) in the plasma as an oxidative stress marker measured by means of Will's method expressed in nmol/ml plasma unit
plasma gluthatione level | eight weeks
  the concentration of glutathione ((2S)-2-Amino-4-{[(1R)-1-[(carboxymethyl)carbamoyl]-2-sulfanylethyl]carbamoyl}butanoic acid) as an endogenous antioxidant compound in the plasma measured by means of Ellman's method expressed in µg/ml plasma unit

SECONDARY OUTCOMES:
days of compliance | eight weeks
  the number of day in which a participant adhere to the assigned dietary plan
mean caloric intake | eight weeks
  the average amount of calories consumed daily by the participant which was determined from food diary and subsequent caloric contents calculation expressed in kilocalorie
mean percentage of caloric intake from protein | eight weeks
  the average proportion of calories obtained from protein compared to the overall daily caloric intake expressed as percentage (%)

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - Civil Workers' Health Service Center of Special Capital Region, Jakarta Pusat, DKI Jakarta
  - Seruni Nutrition Clinic, Jakarta, Jakarta Pusat

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witjaksono F, Jutamulia J, Annisa NG, Prasetya SI, Nurwidya F. Comparison of low calorie high protein and low calorie standard protein diet on waist circumference of adults with visceral obesity and weight cycling. BMC Res Notes. 2018 Sep 21;11(1):674. doi: 10.1186/s13104-018-3781-z. PMID 30241565